CLINICAL TRIAL: NCT04591470
Title: Influence of Inguinal Hernia Repair on Sperm Autoimmunity Using MAR Test
Brief Title: Influence of Inguinal Hernia Repair on Sperm Autoimmunity
Acronym: SPERMAR
Status: Completed | Type: Observational
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: 64/20
Record Dates: First submitted 2020-10-10; First posted 2020-10-19 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-10

CONDITIONS: Male Infertility Due to Antisperm Antibody

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- General population
  Interventions: Diagnostic Test: Mar test
- Pazients undergone inguinal hernia correction
  Interventions: Diagnostic Test: Mar test

INTERVENTIONS:
Diagnostic Test: Mar test — Study of antisperm antibodies

SUMMARY:
Influence of inguinal hernia repair on sperm autoimmunity using MAR test

DETAILED DESCRIPTION:
All infertile male patients, visited between February 2000 and September 2020 and which were tested with MAR (Mixed Autoglobulin Reaction) test, were included in this retrospective study. Sperm quality (number of spermatozoa, motility, vitality and normal forms) were also studied in this patients. The aim of the study is to evaluate if there is a higher incidence of positive MAR test among patients undergoing inguinal hernioplasty compared to the general population

ELIGIBILITY:
Inclusion Criteria:

* Patients undergone to correction of inguinal hernia

Exclusion Criteria:

* No specific exclusion criteria were set.

Ages: 18 Years to 60 Years | Sex: Male
Age Groups: Adult
Study Population: We collected data from all patients who had performed at least one MAR test and a basal spermiogram and who had performed an andrological visit at the Humanitas Clinical Institute in Rozzano (Milan) between February 2000 to September 2020.
Sampling Method: Probability Sample
Enrollment: 2415 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Evaluate if there is a higher incidence of positive MAR test among patients undergoing inguinal hernioplasty | 20 years

SECONDARY OUTCOMES:
Evaluate if there is a modification of seminal parameters among patients undergoing inguinal hernioplasty | 20 years

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Clinico Humanitas, Rozzano, Milano, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gupta S, Krishna A, Jain M, Goyal A, Kumar A, Chaturvedi P, Sagar R, Ramachandran R, Prakash O, Kumar S, Seenu V, Bansal V. A three-arm randomized study to compare sexual functions and fertility indices following open mesh hernioplasty (OMH), laparoscopic totally extra peritoneal (TEP) and transabdominal preperitoneal (TAPP) repair of groin hernia. Surg Endosc. 2021 Jun;35(6):3077-3084. doi: 10.1007/s00464-020-07697-z. Epub 2020 Jun 15. PMID 32556769
- [Background] Stula I, Druzijanic N, Sapunar A, Perko Z, Bosnjak N, Kraljevic D. Antisperm antibodies and testicular blood flow after inguinal hernia mesh repair. Surg Endosc. 2014 Dec;28(12):3413-20. doi: 10.1007/s00464-014-3614-7. Epub 2014 Jun 25. PMID 24962853
- [Background] Matsuda T, Hiura Y, Muguruma K, Okuno H, Horii Y, Yoshida O. Quantitative analysis of testicular histology in patients with vas deferens obstruction caused by childhood inguinal herniorrhaphy: comparison to vasectomized men. J Urol. 1996 Feb;155(2):564-7. PMID 8558661